CLINICAL TRIAL: NCT04561245
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Single and Multiple Ascending Doses of ALT-801 in Healthy Overweight and Obese Volunteers
Brief Title: ALT-801 (Pemvidutide) in Healthy Overweight and Obese Volunteers to Study Safety and Tolerability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-801-101; Pemvidutide (Other: Altimmune)
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Nonalcoholic Steatohepatitis
Keywords: NASH; Obesity
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease | interventions — ALT-801

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ALT-801 (Part 1) (Experimental): Single ascending dose (SAD) cohorts of ALT-801
  Interventions: Drug: ALT-801
- Placebo (Part 1) (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- ALT-801 (Part 2) (Experimental): Multiple ascending dose (MAD) cohorts of ALT-801 administered once weekly for 12 weeks
  Interventions: Drug: ALT-801
- Placebo (Part 2) (Placebo Comparator): Placebo administered once weekly for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ALT-801 — Injected subcutaneously (SC)
  Other Names: Pemvidutide
  Arms: ALT-801 (Part 1); ALT-801 (Part 2)
Other: Placebo — Injected subcutaneously (SC)
  Arms: Placebo (Part 1); Placebo (Part 2)

SUMMARY:
This study was a FIH, Phase 1, randomized, double-blind, placebo-controlled, 2-part single-ascending dose (SAD) and multiple-ascending dose (MAD) study of ALT-801 (pemvidutide) in healthy overweight and obese subjects.

The purpose of the study was to assess the safety and tolerability in healthy overweight and obese volunteers administered single or multiple repeated doses of ALT-801 (pemvidutide).

DETAILED DESCRIPTION:
This study had 2 parts. Part 1 involved single dose cohorts of ALT-801 (pemvidutide) or placebo taken as a subcutaneous (SC) injection and was approximately 36 days in duration. Part 2 involved multiple dose cohorts of ALT-801 (pemvidutide) or placebo taken once a week for 12 weeks as a SC injection and was approximately 116 days in duration. Each participant enrolled in only one part.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers, age 18 to 60 years, inclusive
* Overweight to obese (BMI 25.0 - 40.0 kg/m2)
* MRI-PDFF≥ 10% (Part 2 only)
* Non-smokers or ex-smokers (must have ceased smoking > 1 months prior to screening visit)
* Subjects must otherwise be in good general health, with no significant medical history, have no clinically significant abnormalities on physical examination at screening, and/or before administration of the initial dose of study medication
* Ability and willingness to attend the necessary visits to the study center
* Written informed consent signed prior to entry into the study

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* History of pancreatitis
* History of or acute significant GI disorder
* History of diabetes or use of medications for the treatment of diabetes, or hyperglycemia or HbA1c ≥ 6.5%
* History of clinically significant endocrine (eg, hypothyroidism), neurological, GI, cardiovascular (except controlled hypertension and hypercholesterolemia), hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of neoplastic disease, or personal or family history of multiple endocrine neoplasia or medullary cancer of the thyroid, with the following exceptions:

  1. Adequately treated non-melanomatous skin carcinoma
  2. Female with a history of benign cervical neoplasia if the subject has been compliant with surveillance and treatment as recommended by her physician
* Blood pressure > 150/90 mmHg or heart rate > 100 beats per minute at screening and at Day -1
* Clinically significant laboratory abnormalities including:

Impaired renal function (estimated glomerular filtration rate [eGFR] <60 mL/min/1.73m2) as estimated using the MDRD equation at screening:

1. GFR (mL/min/1.73 m²) = 175 × (SCr/88.4)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American) (SI units), where SCr is standardized serum creatinine in SI units (µmol/L) and age is in years
2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) laboratory values > 2 × upper normal limits
3. Calcitonin > 50 ng/L - Excessive alcohol consumption defined as >21 alcohol units per week for males and as >14 alcohol units per week for females (where 1 unit = half pint of beer, 25 mL of 40% spirit, or 125 mL of wine)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
The Number of Participants with One or More Treatment-Emergent Adverse Events (TEAEs) | Part 1 SAD Cohorts: up to Day 26; Part 2 MAD Cohorts: up to Day 42
Pharmacokinetic (PK): Maximum observed concentration (Cmax) of ALT-801 | Baseline, Day 26
Pharmacokinetic (PK): Area Under the Concentration (AUC) vs Time Curve of ALT-801 | Baseline to Day 26
Change in body weight | Baseline to Week 6
Pharmacodynamic (PD): Change from baseline in magnetic resonance derived proton density fat fraction (MRI-PDFF) | Baseline to Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Altimmune Chief Medical Officer, Study Director — Altimmune, Inc.
Locations (1):
- Nucleus Networks, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No